CLINICAL TRIAL: NCT05767112
Title: Pharmacokinetic Profile of the Calcium-salt and Free Acid Forms of β-hydroxy-β-methylbutyrate in Humans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: HMB pharmacokinetics
Record Dates: First submitted 2023-02-16; First posted 2023-03-14 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Crossover Assignment The order of treatments was be randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HMB-Ca in water (Active Comparator): Investigate whether the pharmacological form of HMB has any impact on its bioavailability and pharmacokinetic profile.
  Interventions: Other: Supplement administation
- HMB-Ca in capsules (Experimental): Avaliate AUC of HMB-Calcium form supplementation.
  Interventions: Other: Supplement administation
- HMB-FA (Experimental): Avaliate AUC of HMB-free acid form supplementation.
  Interventions: Other: Supplement administation

INTERVENTIONS:
Other: Supplement administation — HMB was administred in 3 different forms: 1) HMB-FA in clear capsules; 2) HMB-Ca in gelatine capsules; 3) HMB-Ca dissolved in water. All treatments provided 1g of HMB. Blood samples were taken before and on multiple time points following ingestion.

SUMMARY:
HMB supplementation has been shown to have potential to optimize resistance training responses, which may have important implications for sport, exercise, and health. However, HMB literature shows uncertainties as to which is the superior pharmaceutical form of supplemental HMB (i.e., the calcium salt or the free acid form) in terms of pharmacokinetic profile and bioavailability when consumed by humans. This research project investigated the bioavailability and pharmacokinetics of two different forms of supplemental HMB, namely HMB calcium-salt (HMB-Ca) and HMB Free Acid (HMB-FA). Further, HMB-Ca was provided both diluted in water and encapsulated in gelatine capsules. This pharmacokinetics study adopted a crossover design, open-label design in which male and female participants visited the laboratory on 3 different occasions to receive one the 3 treatments: 1g of HMB; the equivalent of 1g of HMB-Ca in water; the equivalent of 1g of HMB-Ca in gelatine capsules. Venous blood samples were collected before and multiple time points after treatment ingestion, for a period of 12 hours in total. A pre-ingestion midstream urine sample was collected as well as a 24-h post-ingestion total urine sample. All plasma and urine samples were analysed for their HMB concentrations via LC/MS. Time to peak, maximum concentration, area under the curve, half-life time and slope of the incremental phase were calculated to examine the pharmacokinetic profile of HMB and compare the 3 different pharmaceutical forms.

DETAILED DESCRIPTION:
This study aimed to investigate whether the different pharmaceutical forms of HMB show distinct bioavailability and pharmacokinetic profile in humans. A counterbalanced crossover open-label study was conducted. 20 male and female participants were recruited, of which 18 met the inclusion criteria and 16 enrolled in the study. All participants visited the laboratory on 3 different occasions, 5-7 days apart to receive one of the following treatments: 1) 1 g of HMB-FA, or 2) HMB-Ca (equivalent of 1 g of HMB) in capsules, or 3) HMB-Ca (equivalent of 1 g of HMB) dissolved in water. The order of treatments was counterbalanced to control for carryover and order effects using a 3-by-6 (treatment-by-participant) Latin square table (www.statpages.info/latinsq.html). To randomly allocate participants to treatment sequences, participants were recruited in blocks of 6, each containing 3 males and 3 females so that sexes were counterbalanced too. The allocation sequence within each block was defined using a random sequence generator (www.random.org). Blood samples were collected before HBM ingestion and 15, 30, 45, 60, 90, 120, 180, 240, 360 and 720 minutes after HMB ingestion. Urine samples were collected before HMB ingestion (midstream sample) and 24 hours post ingestion (24h total urine). A standardised breakfast was provided to all participants 1h before treatment ingestion. A standardised snack was given to all participants 4 hours after treatment ingestion, and a standardised meal was given 6 hours after treatment ingestion. Water ingestion was standardised in the first 360 minutes after ingestion. In the last 6 hours of the protocol, the participants were dismissed from the lab and returned for the 720 post-ingestion blood collection. They consumed food and water ad-libitum. HMB concentrations were determined in urine and plasma samples by LC/MS using tandem electrospray ionization (ESI). The following pharmacokinetic parameters were calculated: Time to peak, maximum concentration, area under the curve, half-life time and slope of the incremental phase. Plasma and urine HMB concentrations were compared between treatments across time with a 2-factor mixed models analysis. Fixed factors were treatment and time, and participants were the random factor. All pairwise comparisons were adjusted with the Tukey-Kraemer correction. AUC, relative bioavailability, Cmax and Tmax were compared between treatments with repeated measures one-way ANOVA with post-hoc tests adjusted for multiple comparisons using the Bonferroni correction.

ELIGIBILITY:
Inclusion Criteria:

1. age between 18-35 years;
2. ≥150 min of moderate to intense physical activity per week

Exclusion Criteria.

1. smoking,
2. use of statins, anti-inflammatory, or any other medications that could affect lipid metabolism or blood parameters;
3. current or past use of androgenic anabolic steroids;
4. diagnosis of gastric or intestinal disorders that could affect nutrient absorption;
5. diagnosis of kidney or liver disorders that could affect nutrient metabolisation and elimination;
6. any other condition that could be perceived as a potential confounding factor or that could prevent participation in the study.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2016-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Plasma HMB concentration | Up to 720 minutes
  Blood samples collected before and multiple times after treatment ingestion for later determination of plasma HMB concentrations

SECONDARY OUTCOMES:
Urine HMB | Up to 24 hours
  Pre ingestion mid-stream urine sample and 24 hours post ingestion urine

CONTACTS AND LOCATIONS:
Overall Officials: Heitor R Ribeiro, Bsc, Principal Investigator — University of Sao Paulo
Locations (1):
- School of Physical Education and Sport - USP, São Paulo, Brazil